CLINICAL TRIAL: NCT04512677
Title: Ventilatory Weaning Guided by the Timed Inspiratory Effort Index
Brief Title: Ventilatory Weaning Guided by a New Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Timed Inspiratory Effort Index
Record Dates: First submitted 2020-05-28; First posted 2020-08-13 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Respiration, Artificial
Keywords: Mechanical Ventilator; Ventilator Weaning; Spontaneous Breath Test; Predictive Index
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: The secret will be kept by the data collecting investigators and will only be revealed at the end of the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Interventions: Control (No Intervention): Conventional clinical treatment and using the ventilatory weaning protocol and standard extubation with the spontaneous breathing test (SBT) with the T-piece in 30 minutes.
- Experimental: Intervention (Experimental): Conventional clinical treatment and using the Timed Inspiratory Effort (TIE index), which guided the decision to ventilate weaning and extubation.
  Interventions: Device: Timed Inspiratory Effort (TIE index)

INTERVENTIONS:
Device: Timed Inspiratory Effort (TIE index) — Conventional clinical treatment and using the Timed Inspiratory Effort (TIE index), which guided the decision to ventilate weaning and extubation.
  Arms: Experimental: Intervention

SUMMARY:
Mechanical ventilation (MV) is an essential therapy for patients with acute respiratory failure. The ventilatory weaning process should be started when the precipitating causes of the use of the ventilatory prosthesis are resolved. Inappropriately slow weaning exposes the patient to unnecessary discomfort, increases the risk of complications and increases the cost of hospital treatment. In this sense, indices that can predict successful weaning are of great value.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is an essential therapy for patients with acute respiratory failure. The ventilatory weaning process should be started when the precipitating causes of the use of the ventilatory prosthesis are resolved. Inappropriately slow weaning exposes the patient to unnecessary discomfort, increases the risk of complications and increases the cost of hospital treatment. In this sense, indices that can predict successful weaning are of great value. Our study aimed to evaluate the performance of a new ventilatory weaning index, the timed inspiratory effort index (TIE index), as a weaning predictor in comparison with the traditionally used spontaneous breathing test (SBT). The study is a randomized controlled trial of a cohort of mechanically ventilated patients over 24 hours admitted to the ICU of Hospital e Clínica São Gonçalo (HCSG), located in the city of São Gonçalo, State of Rio de Janeiro, Brazil. The TIE index is calculated as the ratio of the maximum inspiratory pressure developed in the last 30 seconds of a 60 second period of unidirectional airway occlusion by the time required to reach this value.

ELIGIBILITY:
Inclusion and exclusion criteria

Our study included patients over 18 years old, under mechanical ventilation, who remained for more than 24 hours of invasive ventilatory assistance and who were able to start the process of weaning. Exclusion criteria comprised tracheostomy, chronic neurological disorders, low level of alertness, and chronic immune suppression states, including positive serology for HIV.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Sucessful weaning | Two years
  Compare the timed inspiratory effort index parameter TIE as an indicator of weaning compared to the spontaneous breathing test

SECONDARY OUTCOMES:
Frequency of failure at weaning | Two years
  Compare the frequency of failure at weaning when using the TIE index or the T-piece TRE as a criterion for extubation.
Counting of the number of tests needed until extubation | Two years
  Evaluate the number of tests required until the decision favorable to extubation was made in both groups.
Comparison of the length of stay in the ICU | Two years
  Compare the length of stay in the ICU between extubation, discharge or death counted from extubation among patients who used the TIE or SBT index in T piece.

OTHER OUTCOMES:
Mortality rate | Two years
  Compare the ICU mortality among patients using the TIE or TRE method in T piece

CONTACTS AND LOCATIONS:
Overall Officials: Jecemir R Lugon, MD, PhD, Principal Investigator — Universidade Federal Fluminense; Marcos p Godoy, PT, MSc, Study Chair — Hospital e Clínica São Gonçalo
Locations (2):
- Brazil (2):
  - Universidade Federal Fluminense, Niterói, Rio de Janeiro
  - Hospital e Clínica São Gonçalo, São Gonçalo, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacIntyre N. Another Look at Outcomes from Mechanical Ventilation. Am J Respir Crit Care Med. 2017 Mar 15;195(6):710-711. doi: 10.1164/rccm.201610-1988ED. No abstract available. PMID 28294658
- [Result] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Result] de Souza LC, Guimaraes FS, Lugon JR. Evaluation of a new index of mechanical ventilation weaning: the timed inspiratory effort. J Intensive Care Med. 2015 Jan;30(1):37-43. doi: 10.1177/0885066613483265. Epub 2013 Apr 10. PMID 23753238
- [Result] da Silva Guimaraes B, de Souza LC, Cordeiro HF, Regis TL, Leite CA, Puga FP, Alvim SH, Lugon JR. Inspiratory Muscle Training With an Electronic Resistive Loading Device Improves Prolonged Weaning Outcomes in a Randomized Controlled Trial. Crit Care Med. 2021 Apr 1;49(4):589-597. doi: 10.1097/CCM.0000000000004787. PMID 33332819
- [Result] da Silva Guimaraes BL, de Souza LC, Guimaraes FS, Lugon JR. Serial Weekly Measurements of the Timed Inspiratory Effort Index Can Predict Successful Prolonged Weaning. Respir Care. 2019 Oct;64(10):1286-1292. doi: 10.4187/respcare.06367. Epub 2019 Mar 26. PMID 30914494
- [Result] de Souza LC, Guimaraes FS, Lugon JR. The timed inspiratory effort: a promising index of mechanical ventilation weaning for patients with neurologic or neuromuscular diseases. Respir Care. 2015 Feb;60(2):231-8. doi: 10.4187/respcare.03393. Epub 2014 Oct 28. PMID 25352688
- [Result] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Result] Subira C, Hernandez G, Vazquez A, Rodriguez-Garcia R, Gonzalez-Castro A, Garcia C, Rubio O, Ventura L, Lopez A, de la Torre MC, Keough E, Arauzo V, Hermosa C, Sanchez C, Tizon A, Tenza E, Laborda C, Cabanes S, Lacueva V, Del Mar Fernandez M, Arnau A, Fernandez R. Effect of Pressure Support vs T-Piece Ventilation Strategies During Spontaneous Breathing Trials on Successful Extubation Among Patients Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2019 Jun 11;321(22):2175-2182. doi: 10.1001/jama.2019.7234. PMID 31184740
- [Result] Sklar MC, Burns K, Rittayamai N, Lanys A, Rauseo M, Chen L, Dres M, Chen GQ, Goligher EC, Adhikari NKJ, Brochard L, Friedrich JO. Effort to Breathe with Various Spontaneous Breathing Trial Techniques. A Physiologic Meta-analysis. Am J Respir Crit Care Med. 2017 Jun 1;195(11):1477-1485. doi: 10.1164/rccm.201607-1338OC. PMID 27768396
- [Result] Girard TD, Alhazzani W, Kress JP, Ouellette DR, Schmidt GA, Truwit JD, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Morris PE; ATS/CHEST Ad Hoc Committee on Liberation from Mechanical Ventilation in Adults. An Official American Thoracic Society/American College of Chest Physicians Clinical Practice Guideline: Liberation from Mechanical Ventilation in Critically Ill Adults. Rehabilitation Protocols, Ventilator Liberation Protocols, and Cuff Leak Tests. Am J Respir Crit Care Med. 2017 Jan 1;195(1):120-133. doi: 10.1164/rccm.201610-2075ST. PMID 27762595
- [Result] Jung B, Moury PH, Mahul M, de Jong A, Galia F, Prades A, Albaladejo P, Chanques G, Molinari N, Jaber S. Diaphragmatic dysfunction in patients with ICU-acquired weakness and its impact on extubation failure. Intensive Care Med. 2016 May;42(5):853-861. doi: 10.1007/s00134-015-4125-2. Epub 2015 Nov 16. PMID 26572511